CLINICAL TRIAL: NCT02261831
Title: Identify Bacteria Associated With Metabolic Diseases That Reside Both in Intestinal Crypts and in Blood.
Acronym: MICIMAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13 6936 03
Record Dates: First submitted 2014-07-22; First posted 2014-10-10 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Obesity
Keywords: bacterial; gut; type 2 diabetes.; 16S rDNA gene; intestinal crypt
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- obese patients (Experimental): Total blood sample, and 4 biopsies : collection of 2 colonic and 2 ileal biopsies
  Interventions: Other: obese patients
- Diabetic patients (Experimental): Total blood sample, and 4 biopsies : collection of 2 colonic and 2 ileal biopsies
  Interventions: Other: diabetic patients
- Patients free of obesity and diabetes (Experimental): Total blood sample, and 4 biopsies : collection of 2 colonic and 2 ileal biopsies
  Interventions: Other: patients free of obesity and diabetes
- patients free type 2 diabetes. (Experimental): Total blood sample, and 4 biopsies : collection of 2 colonic and 2 ileal biopsies
  Interventions: Other: patients free type 2 diabetes

INTERVENTIONS:
Other: obese patients — collection of blood sampling and biopsies
  Arms: obese patients
Other: diabetic patients — collection of blood sampling and biopsies
  Arms: Diabetic patients
Other: patients free of obesity and diabetes — collection of blood sampling and biopsies
  Arms: Patients free of obesity and diabetes
Other: patients free type 2 diabetes — collection of blood sampling and biopsies
  Arms: patients free type 2 diabetes.

SUMMARY:
The investigators will compare 16sRDNA profile in cases and controls in order to identify bacteria associated with metabolic diseases that reside both in intestinal crypts and in blood.

DETAILED DESCRIPTION:
Experimental evidence suggests that bacterial translocation from gut to tissue could be an initial step leading to diabetes. To test this hypothesis, a bacterial component that is highly conserved between different species of bacteria, the 16S rDNA gene will be analysed both in intestinal crypt and in blood in patients with type 2 diabetes, obese patients and control.

ELIGIBILITY:
Inclusion Criteria:

* Between 35 and 75 years old
* Colonoscopy and biopsies required

Diabetes population:

* Type 2 diabetes

Obese population:

* Android obesity

Exclusion Criteria:

* Inflammatory bowel disease
* Colonic cancer
* Bariatric surgery
* Previous administration of antibiotic (within 15 days)
* Pregnancy

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2014-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
rDNA comparison between cases and controls | 36 months
  Comparison of 16sRDNA profile in cases and controls in order to identify bacteria associated with metabolic diseases that reside both in intestinal crypts and in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques AMAR, MD PhD, Study Director — University Hospital, Toulouse; Jacques Moreau, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France